CLINICAL TRIAL: NCT00003761
Title: A Phase I Trial of Recombinant Vaccinia Virus That Expresses DF3/MUC1 in Patients With Metastatic Adenocarcinoma of the Breast
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Donald W. Kufe, Kufe, Donald William,M.D., Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-050; U01CA062490 (NIH); P30CA006516 (NIH); NCI-T98-0057 (Other: Protocol relative to DFPCC #97-050)
Record Dates: First submitted 1999-11-01; First posted 2003-12-10 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rV-DF3/MUC1 (Experimental): * rV-DF3/MUC1 vaccinations will be administered 4 week intervals for a total of 3 doses.
  * Participants will be followed weekly until 28 days after the final dose (day 85) then month for 6 months
  Interventions: Biological: rV-DF3/MUC1

INTERVENTIONS:
Biological: rV-DF3/MUC1 — - The starting dose for this Phase I study of rV-DF3/MUC1 will be 4.76 x 106 PFU.
  -- Dose escalation will proceed with cohorts of at least 6 patients as follows: Per vaccination
  * Level 1 4.76 x 106 PFU
  * Level 2 4.76 x 107 PFU
  * Level 3 4.76 x 108 PFU

SUMMARY:
This protocol is designed to evaluate the side effects of rV-DF3/MUC1 and to determine the safest dose which should be used in the treatment of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity associated with repeated vaccination with recombinant vaccinia DF3/MUC1 vaccine (rV-DF3/MUC1) in patients with metastatic breast cancer. II. Determine the maximum tolerated dose of rV-DF3/MUC1, based on cellular and humoral immunity, in these patients. III. Determine whether vaccination with rV-DF3/MUC1 is associated with antitumor activity in these patients.

OUTLINE: This is an open label, dose escalation study. Patients receive recombinant vaccinia DF3/MUC1 vaccine (rV-DF3/MUC1) intradermally. Treatment repeats every month for 3 courses in the absence of disease progression or unacceptable toxicity. Cohorts of at least 6 patients receive escalating doses of rV-DF3/MUC1 until the maximum tolerated dose (MTD) or the highest dose level to be tested is reached. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed monthly for 6 months.

PROJECTED ACCRUAL: A total of 16-28 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
* Inclusion Criteria
* Patients with a histologically confirmed diagnosis of metastatic adenocarcinoma of the breast. Patients may have measurable disease, but it is not required. Patients may have received any number of prior therapies for metastatic disease. Untreated patients are also eligible.
* Age ≥ 18 years
* Patients must have an ECOG = Performance Status of 0-1
* Patients must have a WBC > 2000/mm 3 and a platelet count > 100,000/mm3.
* Patients must have adequate renal function documented by a serum creatinine < 2.0 mg/d1.
* Patients must have adequate liver function demonstrated by a serum bilirubin < 2.0 mg/di, and a SGPT < 4 times the upper limit of normal.
* ≥3 weeks since chemotherapy (> 6 weeks for nitosoureas or mitomycin C), hormonal therapy or radiation therapy
* Immunologic testing must be at least normal as defined by at least normal delayed type hypersensitivity, at least normal CD4: CD8 ratio (>1), at least normal lymphocyte proliferation testing (to Con A), and at least normal immunoglobulin levels
* Patients must not have evidence of altered immune responsiveness or autoimmune syndromes (scleroderma,systemic lupus erythematosus, etc.). Patients must be HIV negative. This treatment may be associated with increased adverse effects for individuals with immune deficiencies, and HIV-associated symptoms preclude accurate assessment of toxicity.
* Patients must not have undergone splenectomy.
* Patients with active cases or history of extensive skin disorders (such as extensive psoriasis, burns, impetigo, disseminated zoster) are ineligible.
* Patients must not have any other serious medical condition which in the opinion of the investigator is incompatible with the protocol. Patients with active infections requiring antibiotics are not eligible until the infection has cleared and the antibiotics have been stopped for at least 3 days.
* Patients must be able to avoid close contact with children < 3 years of age, pregnant women, individuals with eczema or skin conditions and immune suppressed individuals during a period of two weeks after each vaccination.
* Patients must have had prior vaccinia (small pox) exposure.
* Tumor tissue positive for staining with MAbs DF3 and/or DF3-P or elevated serum CA15-3. Note: This can be done on stored slides.
* Patients must not have a history of seizures, encephalitis or multiple sclerosis.
* Patients must not be allergic to eggs.
* Patients must not be pregnant or breast-feeding due to a possible increased risk with exposure to vaccinia virus of both mother and newborn as well as unknown risks to the fetus.
* Signed informed consent.
* Exclusion Criteria
* Patients must not have evidence of altered immune responsiveness or autoimmune syndromes (scleroderma, systemic lupus erythematosus, etc.). Patients must be HIV negative This treatment may be associated with increased adverse effects for individuals with immune deficiencies, and HIV-associated symptoms preclude accurate assessment of toxicity.
* Patients must not have undergone splenectomy
* Patients with active cases or history of extensive skin disorders (such as extensive psoriasis, burns, impetigo, disseminated zoster) are ineligible.
* Patients must not have any other serious medical condition which in the opinion of the investigator is incompatible with the protocol. Patients with active infections requiring antibiotics are not eligible until the infection has cleared and the antibiotics have been stopped for at least 3 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1999-03-03 (Actual); Primary Completion 2001-04-20 (Actual); Study Completion 2001-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald W. Kufe, MD, Study Chair — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No